CLINICAL TRIAL: NCT04781309
Title: A Pilot Study of NT-I7, a Long-Acting Recombinant IL-7 Molecule, as an Immune Reconstitution Strategy for Lymphopenia in Patients With Progressive Multifocal Leukoencephalopathy
Brief Title: NT-I7, a Long-Acting Recombinant IL-7 Molecule, as an Immune Reconstitution Strategy for Lymphopenia in Patients With Progressive Multifocal Leukoencephalopathy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: NeoImmuneTech (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000126; 000126-N
Record Dates: First submitted 2021-03-03; First posted 2021-03-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11-14

CONDITIONS: Progressive Multifocal Leukoencephalopathy
Keywords: Absolute Lymphocyte Count; safety and tolerability of NT-I7
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal | interventions — efineptakin alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NT-I7 (Experimental): 480 microgram/kg IM (initial dose)
  Interventions: Drug: NT-I7

INTERVENTIONS:
Drug: NT-I7 — NT-I7 is a recombinant human interleukin-7 fused to a hybrid fragment crystallizable region of a human antibody (hyFc). NT-I6 has a molecular weight of 104 kD. The active moiety of NT-I7 is recombinant human interleukin-7 (rhIL-7), containing human IL-7 (amino acids 4 through 155) and exhibiting all known functions of endogenous human IL-7.

SUMMARY:
Background:

Progressive multifocal leukoencephalopathy (PML) is a brain infection. It is caused by a virus. PML can happen in people with a weakened immune system. PML is associated with cognitive and visual impairment as well as motor and speech disturbances. There is no treatment for PML. Researchers want to see if a new drug can help.

Objective:

To see if the drug NT-I7 can help increase lymphocyte numbers, which may help control PML infection.

Eligibility:

Adults ages 18 and older with PML who are enrolled in Protocol #13-N-0017.

Design:

Participants will be screened under Protocol #13-N-0017.

Participants will have a 7-day inpatient stay, outpatient visits, and follow-up phone calls.

Participants will have a medical history and physical exam. They will give urine samples. Blood will be drawn from an arm vein or through an intravenous (IV) catheter.

Participants will get up to 3 doses of NT-I7. It will be given by injection into the muscle.

Participants will have lumbar punctures ( spinal taps ). A thin needle will be inserted into the spinal canal in the lower back. Cerebrospinal fluid will be removed. X-ray may be used to guide the procedure.

Participants will have magnetic resonance imaging (MRI) of the brain. The MRI scanner is a metal cylinder surrounded by a magnetic field. During MRIs, participants will lie on a table that slides in and out of the scanner. Soft padding or a coil will be placed around their head. They will get gadolinium, a contrast agent, through an IV catheter.

Participation will last for 12 to 19 months.

...

DETAILED DESCRIPTION:
Study Description:

This protocol will test whether NT-I7 is a viable strategy for promoting immune reconstitution in lymphopenic patients with PML. Twelve evaluable adults with PML and lymphopenia (CD4 or CD8 T cell count of <=200 cells/dL), without a history of autoimmune disease affecting vital organs, will complete this pilot study. Patients will be observed as inpatient for the first 7 days following any experimental drug dosing. To follow, patients will return to NIH for a second 7-day inpatient stay by Day 21, and then for scheduled outpatient visits at NIH at month 2, 3, 6, 9 and 12 following any drug dosing. Follow up phone calls will be conducted at month 4, 5, 7 and 8. Patients may be eligible for a second dose of NT-I7 at higher dose if target ALC (1000/microliter) not reached, or at same dose if initial response is adequate but not sustained, for a maximum of 3 doses. The primary outcome measure is change in absolute lymphocyte counts (ALC). Secondary outcomes include safety and tolerability. Exploratory clinical, radiological, and laboratory measures will be obtained to investigate mechanism of action of NT-I7 and for biomarker development.

Objectives:

Primary Objective: To determine the kinetics and magnitude of effect of NT-I7 on absolute lymphocyte counts in patients with PML and underlying lymphopenia from various causes, in order to inform appropriate design of a future study.

Secondary Objectives: (1) To assess safety and tolerability of NT-I7. (2) To determine kinetics and magnitude of effect of NT-I7 on lymphocyte subsets. (3) To investigate effect of NT-I7 on PML disease course. (4) To investigate mechanism of action of NT-I7.

Endpoints:

Primary Endpoint: Change in absolute lymphocyte counts (ALC) over 6 months.

Secondary Endpoints: (1) Adverse event tables. (2) Change in lymphocyte subset counts, including CD4, CD8 and CD19 positive cells (3) Change in standardized disability rating scales, PML lesion extension by brain MRI, viral quantification in CSF and survival. (4) Exploratory serological and CSF measures to investigate immune response to JCV and mechanism of action of NT-I7.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults (18 years of age or older)
* Definite or Probable PML (2013 AAN Consensus Diagnostic Criteria)
* CD4 and/or CD8 lymphopenia <= 200 cells/dL that is not readily reversible within one month
* Enrolled in 13-N-0017
* Ability to provide own consent at study entry
* Ability to travel to NIH for study visits
* Willingness to comply with all study procedures
* If able to become pregnant or to father a child, patient must agree to commit to the use of a reliable/accepted method of birth control (i.e. hormonal contraception (birth control pills, injected hormones, vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or surgical sterilization (hysterectomy, tubal ligation, or vasectomy) for the duration of the study

EXCLUSION CRITERIA:

* Age < 18 years of age
* Ongoing treatment with immune-suppressive medications (exception: topical steroid use and all forms of systemic steroids with durations less than 2 weeks)
* History of immune-mediated disease affecting vital organ
* Concurrent treatment with experimental therapies for PML that would interfere with or confound assessment of study outcomes
* History of underlying autoimmune disease involving the CNS
* Contraindication to any study procedures that would compromise ability to safely monitor the patient
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial or interfere with study participation; or not in the best interest of the subject to participate, in the opinion of the treating investigator
* Women who are pregnant or breastfeeding
* Unwilling to have coded samples and/or data saved or used in other studies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
the longitudinal change in absolute lymphocyte count over 6 months following study drug administration | over 6months following study drug administration
  determine the kinetics and magnitude of effect of NT-I7 on absolute lymphocyte counts (ALC) in patients with PML and underlying lymphopenia from various causes, in order to inform appropriate design of a future study

SECONDARY OUTCOMES:
Safety | at each study timepoint
  assessed by the occurrence of treatment-related adverse events. These adverse events will be tabulated separately by timepoint to identify any trends in the data and will be described using number and percent.
Change in lymphocyte subsets, including CD4, CD8, and CD19 positive cells | at each study timepoint
  These values will be investigated first descriptively at each timepoint using mean and SD or median and IQR, and then graphically. Key comparisons of interest will include baseline to Month 3 and baseline to Month 6.
Disease course | at each study timepoint
  These endpoints include quantification of JCV DNA in CSF and blood, change in Modified Rankin Scale score, change in Karnofsky Performance Scale score, change in PML lesion extension, change in pattern of contrast enhancement by brain MRI and survival. Key comparisons of interest will include baseline to Month 3 and baseline to Month 6. Here, the goal is to provide some initial proof of principle that the disease course is being impacted in a measurable way, particularly beyond Month 3.

CONTACTS AND LOCATIONS:
Overall Officials: Irene CM Cortese, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000126-N.html